CLINICAL TRIAL: NCT01387178
Title: Outcomes From Initial Maintenance Therapy With Fluticasone Propionate 250/Salmeterol 50 (FSC) or Tiotropium in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111267
Record Dates: First submitted 2011-06-16; First posted 2011-07-04 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: chronic obstructive pulmonary disease; cost and cost analysis; bronchodilators; healthcare utilization; fluticasone propionate/salmeterol; tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination; Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD patients - risk analysis population: Patient-records from patients aged 40 and older with at least 2 medical claims with a diagnosis of COPD, at least on diagnosis in the 12 months prior to the index date and at least one diagnosis in the post-index date observation period, and at least one prescription claim for either FSC 250 µg/50µg or TIO. Patient records for the risk analysis population will be required to have continuous medical and pharmacy health plan enrollment for at least 12 months before and at least 3 months after the index date. The index date will be defined as the date of the first prescription claim for FSC or TIO (between January 1, 2004 and June 30, 2008).
  Interventions: Drug: fluticasone propionate/salmeterol 250µg/50µg (FSC); Drug: tiotropium bromide (TIO)
- COPD patients - cost analysis population: Patient-records from patients aged 40 and older with at least 2 medical claims with a diagnosis of COPD, at least on diagnosis in the 12 months prior to the index date and at least one diagnosis in the post-index date observation period, and at least one prescription claim for either FSC 250 µg/50µg or TIO. The cost analysis population is a subset of the risk analysis population. Patient records for the cost analysis population will be required to have continuous medical and pharmacy health plan enrollment for at least 12 months before and at least 12 months after the index date. The index date will be defined as the date of the first prescription claim for FSC or TIO (between January 1, 2004 and September 30, 2007).
  Interventions: Drug: fluticasone propionate/salmeterol 250µg/50µg (FSC); Drug: tiotropium bromide (TIO)

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol 250µg/50µg (FSC) — Patient records with evidence of COPD and prescription claims for FSC
  Other Names: Advair®
Drug: tiotropium bromide (TIO) — Patient records with evidence of COPD and prescription claims for TIO
  Other Names: Spriva®

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by chronic airflow limitation caused by inflammation-mediated damage to lung tissue. Although damage to lung tissue in COPD appears to be irreversible, evidence suggests that the course of COPD can be altered through measures such as smoking cessation, pulmonary rehabilitation, and the use of pharmacotherapy for bronchodilation. A primary goal of maintenance pharmacotherapy is to reduce the incidence of acute exacerbations and the associated hospitalizations and emergency department (ED) visits. Bronchodilation in COPD maintenance therapy can be accomplished with the long-acting anticholinergic tiotropium (TIO), long acting beta-agonists (e.g. formoterol, salmeterol), methylxanthines (e.g. theophylline), or combination therapy with a long-acting beta-agonist and an inhaled corticosteroid (e.g. fluticasone propionate/salmeterol [FSC]).

The objective of this study is to compare the benefits of combination long-acting beta-agonist/inhaled corticosteroid therapy to long-acting anticholinergic therapy. The study compares the risk of COPD exacerbations and COPD-related healthcare utilization and costs for commercially-insured patients age 40 and older who were prescribed FSC to those prescribed TIO. The null hypothesis is that no difference exists between the costs and outcomes of COPD patients treated with TIO and those treated with FSC. The test hypothesis is that patients treated with either TIO or FSC will incur lower costs and use fewer healthcare resources for the management of COPD.

The source of data for this study was the Ingenix Impact database (formerly the Integrated Healthcare Information Services [IHCIS] database). This is an administrative claims database that includes patient-level data on enrollment, facility, professional, and pharmacy services from approximately 50 million patients covered by more than 40 managed care health plans across the United States (US).

The study design is a retrospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is age 40 or older
* Patient record indicates a new prescription claim for fluticasone propionate/salmeterol (FSC) or tiotropium bromide (TIO) (first pharmacy claim defines the index date)
* Patient records include at least two medical claims with a primary or non-primary diagnosis of COPD (International Classification of Disease-9 [ICD-9] code 490.xx - 492.xx or 496.xx)
* At least one of the patient's ICD-9 codes for COPD is observed in the 12 months prior to the first pharmacy claim for FSC or TIO (the index date)

Exclusion Criteria:

* A pharmacy claim for FSC or TIO prior to the index date
* The patient initiated FSC at a dose other than 250µg/50µg
* The patient initiated FSC and TIO at the same time
* The patient had one or more prescription with missing dosing information
* The patient had a prescription claim for the study medication other than the one they started on at the index date within 60 days after the index date

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient records for commercially-insured patients with chronic obstructive pulmonary disease (COPD) aged 40 and older. For the risk-analysis population, patients were required to have at least 12 months of continuous enrollment prior to the index date and at least 3 months of continuous enrollment after the index date. A subgroup analysis was conducted for costs that included patients in the total population who also had at least 12 months of continuous coverage following the index date (the cost-analysis population).
Sampling Method: Non-Probability Sample
Enrollment: 22223 (Actual)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a cohort. All diagnoses and treatments are recorded in the course of routine medical practice.
Groups:
- Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg: Participants 40 years of age or older with >=2 medical claims with a primary or non-primary diagnosis of Chronic Obstructive Pulmonary Disease (COPD) (International Classification of Disease, 9th Edition, Clinical Modification [ICD-9-CM] code 490.xx, 491.xx, 492.xx, or 496.xx), >=1 in the 12 months prior to the index date (defined as the first pharmacy claim for the study drug), >=1 in the post-index date observation period, and >=1 prescription claim for fluticasone/propionate 250 µg /50 µg (FSC)
- Tiotropium Bromide 18 µg: Participants 40 years of age or older with >=2 medical claims with a primary or non-primary diagnosis of COPD (ICD-9-CM code 490.xx, 491.xx, 492.xx, or 496.xx), >=1 in the 12 months prior to the index date (defined as the first pharmacy claim for the study drug), >=1 in the post-index date observation period, and >=1 prescription claim for tiotropium bromide (TIO)
Period: Overall Study
Arm/Group | Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg | Tiotropium Bromide 18 µg
Started | 11582 | 10641
Completed | 11582 | 10641
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg: Participants 40 years of age or older with >=2 medical claims with a primary or non-primary diagnosis of COPD (ICD-9-CM code 490.xx, 491.xx, 492.xx, or 496.xx), >=1 in the 12 months prior to the index date (defined as the first pharmacy claim for the study drug), >=1 in the post-index date observation period, and >=1 prescription claim for FSC
- Tiotropium Bromide 18 µg: Participants 40 years of age or older with >=2 medical claims with a primary or non-primary diagnosis of COPD (ICD-9-CM code 490.xx, 491.xx, 492.xx, or 496.xx), >=1 in the 12 months prior to the index date (defined as the first pharmacy claim for the study drug), >=1 in the post-index date observation period, and >=1 prescription claim for TIO
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg | Tiotropium Bromide 18 µg | Total
Number analyzed (Participants) | 11582 | 10641 | 22223
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (10.6) | 63.1 (10.0) | 61.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6121 | 4958 | 11079
  Male | 5461 | 5683 | 11144
Region of Enrollment [Number; unit: Participants] — Some participants are grouped into the "National" region to protect their identities because the combination of their medical and demographic information is considered "infrequent" and could potentially be used to identify the participants.
  Participants
    Northeast | 4523 | 4149 | 8672
    South | 3818 | 3630 | 7448
    Midwest | 1790 | 1731 | 3521
    West | 1085 | 827 | 1912
    National or Unknown | 366 | 304 | 670
Number of participants with the indicated payer source [Number; unit: participants] — Participants were classified according to the type of healthcare payer with which they were associated.
  participants
    Commercial | 10233 | 9227 | 19460
    Medicaid | 121 | 50 | 171
    Medicare | 1228 | 1364 | 2592
Charlson Comorbidity Score [Mean (Standard Deviation); unit: scores on a scale] — The Charlson Comorbidity Index estimates 10-year mortality risk. Scores range from 0 - 37, with a lower score indicating a higher chance of survival.
  scores on a scale | 1.6 (2.1) | 1.6 (2.2) | 1.6 (2.1)
Number of the Indicated Pre-Index Period COPD-related comorbidities [Number; unit: number of comorbidities] — The pre-index period was defined as the 12 months prior to the index date, which corresponded with the start of the study medication.
  number of comorbidities
    Asthma | 3326 | 1651 | 4977
    Congestive heart failure | 1472 | 1624 | 3096
    Upper respiratory infection | 4395 | 2952 | 7347
    Lower respiratory infection | 531 | 475 | 1006
Number of the Indicated Pre-Index Period Treatments [Number; unit: number of treatments]
  Long-acting beta-agonist use | 242 | 556 | 798
  Oxygen use | 1210 | 1517 | 2727
Number of Participants with the Indicated COPD Severity [Number; unit: participants] — Mild, moderate, and severe COPD were defined by an algorithm for retrospective data analyses that is based on COPD-related healthcare encounters such as intensive care unit stays, hospitalizations, emergency department/urgent care visits, and the use of oxygen.
  participants
    Mild | 9442 | 8476 | 17918
    Moderate | 750 | 520 | 1270
    Severe | 1390 | 1645 | 3035

OUTCOME MEASURES:

1. Primary Outcome: Post-index Period COPD-related, Unadjusted Costs
Description: The mean cost per participant for COPD-related healthcare interventions for one year following the index date (first pharmacy claim for fluticasone propionate/salmeterol 250 µg/50 µg [FSC] or tiotropium bromide [TIO]) was calculated. Total medical costs included inpatient, emergency department, and outpatient costs associated with the treatment of COPD. Total pharmacy costs included costs of all COPD-related medications, and total healthcare costs included all medical and pharmacy costs that were related to COPD treatment. These costs were unadjusted and reflect the actual costs.
Time Frame: 1 year
Population: A subpopulation of participants with an index date between January 1, 2004 and September 30, 2007
Measure: Mean (Standard Deviation); unit: United States (US) dollars
Arm/Group | Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg | Tiotropium Bromide 18 µg
Number analyzed (Participants) | 7933 | 6372
United States (US) dollars
  Inpatient services | 688 (4998) | 867 (6887)
  Emergency department visits | 55 (415) | 52 (363)
  Inpatient and emergency department visits | 743 (5090) | 919 (6977)
  Office visits | 231 (388) | 293 (559)
  Other outpatient/ancillary services | 734 (2504) | 879 (3050)
  Total medical costs | 1709 (6322) | 2091 (8302)
  Total pharmacy costs | 1291 (1791) | 1209 (1378)
  Total healthcare utilization | 3000 (6805) | 3299 (8536)
Statistical Analysis 1: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg; Test type: Superiority or Other; Adjusted Mean = 7451, 95% CI 2-sided [5857 to 9045] — The mean predicted cost for inpatient services for participants treated with FSC. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 2: Comparison: Tiotropium Bromide 18 µg; Test type: Superiority or Other; Adjusted Mean = 11545, 95% CI 2-sided [8827 to 14263] — The mean predicted cost for inpatient services for participants treated with TIO. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 3: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg; Test type: Superiority or Other; Adjusted Mean = 61, 95% CI 2-sided [58 to 63] — The mean predicted cost for emergency department visits for participants treated with FSC. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 4: Comparison: Tiotropium Bromide 18 µg; Test type: Superiority or Other; Adjusted Mean = 51, 95% CI 2-sided [49 to 53] — The mean predicted cost for emergency department visits for participants treated with TIO. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 5: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg; Test type: Superiority or Other; Adjusted Mean = 231, 95% CI 2-sided [227 to 234] — The mean predicted cost for office visits for participants treated with FSC. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 6: Comparison: Tiotropium Bromide 18 µg; Test type: Superiority or Other; Adjusted Mean = 295, 95% CI 2-sided [290 to 299] — The mean predicted cost for office visits for participants treated with TIO. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 7: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg; Test type: Superiority or Other; Adjusted Mean = 873, 95% CI 2-sided [827 to 919] — The mean predicted cost for other outpatient and ancillary services for FSC participants. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 8: Comparison: Tiotropium Bromide 18 µg; Test type: Superiority or Other; Adjusted Mean = 1080, 95% CI 2-sided [1022 to 1138] — The mean predicted cost for other outpatient and ancillary services for TIO participants. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 9: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg; Test type: Superiority or Other; Adjusted Mean = 1267, 95% CI 2-sided [1251 to 1283] — The mean predicted cost for pharmacy services for participants treated with FSC. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 10: Comparison: Tiotropium Bromide 18 µg; Test type: Superiority or Other; Adjusted Mean = 1250, 95% CI 2-sided [1234 to 1266] — The mean predicted cost for pharmacy services for participants treated with TIO. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 11: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg; Test type: Superiority or Other; Adjusted Mean = 1175, 95% CI 2-sided [1083 to 1267] — The mean predicted cost for inpatient and emergency department services for FSC participants. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 12: Comparison: Tiotropium Bromide 18 µg; Test type: Superiority or Other; Adjusted Mean = 1566, 95% CI 2-sided [1438 to 1695] — The mean predicted cost for inpatient and emergency department services for TIO participants. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 13: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg; Test type: Superiority or Other; Adjusted Mean = 2991, 95% CI 2-sided [2922 to 3059] — The mean predicted cost for total healthcare services for participants treated with FSC. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used
Statistical Analysis 14: Comparison: Tiotropium Bromide 18 µg; Test type: Superiority or Other; Adjusted Mean = 3304, 95% CI 2-sided [3221 to 3386] — The mean predicted cost for total healthcare services for participants treated with TIO. A generalized linear model with a log link function and gamma distribution for the error term to resolve the issue of skewed cost distribution was used

2. Primary Outcome: Mean Number of COPD Exacerbations
Description: Moderate COPD exacerbations were defined as the occurrence of a COPD-related emergency department (ED) visit or a COPD-related office visit that is closely followed by a prescription claim for oral steroids or antibiotics. Severe exacerbations were defined as the occurrence of a COPD-related hospital admission.
Time Frame: 1 year
Population: The total population including participants with index dates between January 1,2004 and June 30, 2008.
Measure: Mean (Standard Deviation); unit: number of exacerbations
Arm/Group | Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg | Tiotropium Bromide 18 µg
Number analyzed (Participants) | 11582 | 10641
number of exacerbations
  Moderate Exacerbation | 0.35 (0.77) | 0.29 (0.71)
  Severe Exacerbation | 0.05 (0.29) | 0.05 (0.32)
  Any Exacerbation | 0.4 (0.87) | 0.34 (0.82)
Statistical Analysis 1: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg vs Tiotropium Bromide 18 µg; Test type: Superiority or Other; p = 0.2198, Regression, Cox — Risk of Moderate COPD Exacerbations; Hazard Ratio (HR) = 0.964, 95% CI [0.909 to 1.022]
Statistical Analysis 2: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg vs Tiotropium Bromide 18 µg; Test type: Superiority or Other; p = 0.0406, Regression, Cox — Risk of Severe COPD Exacerbations; Hazard Ratio (HR) = 0.864, 95% CI [0.752 to 0.994]
Statistical Analysis 3: Comparison: Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg vs Tiotropium Bromide 18 µg; Test type: Superiority or Other; p = 0.0962, Regression, Cox — Risk of Any COPD Exacerbation; Hazard Ratio (HR) = 0.953, 95% CI [0.901 to 1.009]

3. Secondary Outcome: Number of COPD-related Healthcare Encounters
Time Frame: 1 year
Population: A subpopulation of participants with an index date between January 1, 2004 and September 30, 2007
Measure: Number; unit: number of encounters
Arm/Group | Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg | Tiotropium Bromide 18 µg
Number analyzed (Participants) | 7933 | 6372
number of encounters
  Inpatient services | 2155 | 1792
  Emergency department visits | 3085 | 2312
  Inpatient and emergency department visits | 3673 | 2817
  Office visits | 7833 | 6295
  Other outpatient/ancillary services | 7243 | 5859

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | Fluticasone Propionate/Salmeterol 250 Micrograms (µg)/50 µg | Tiotropium Bromide 18 µg
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.